CLINICAL TRIAL: NCT00390481
Title: Randomized Evaluation of Carotid Occlusion and Neurocognition (RECON)
Brief Title: Study of Carotid Occlusion and Neurocognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Randolph S. Marshall, Professor at Affil Hosp/Inst, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAA8456; 5R01NS048212 (NIH)
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Carotid Artery Diseases
Keywords: Carotid Occlusion; Cognition
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): EC-IC Bypass
  Interventions: Procedure: EC-IC Bypass in the COSS study
- Control (No Intervention): Best Medical Therapy

INTERVENTIONS:
Procedure: EC-IC Bypass in the COSS study — EC-IC Bypass surgery involves taking an artery from the scalp outside the skull, making a small hole in the skull, and then connecting the scalp artery to a brain artery inside the skull. In this way, the blockage of the carotid artery in the neck is bypassed and more blood can flow to the brain.
  Arms: Intervention

SUMMARY:
To determine the relationship between cognitive functioning and blood flow in the brain among patients randomized to either extracranial-intracranial (EC-IC) bypass or medical therapy alone in the Carotid Occlusion Surgery Study (COSS).

DETAILED DESCRIPTION:
The Carotid Occlusion Surgery Study (COSS) evaluates whether a surgical operation, EC-IC bypass surgery, can reduce the chance of a stroke in someone who has complete blockage in one main artery in the neck that supplies blood to the brain (the carotid artery). The operation bypasses the blockage so more blood can flow to the brain. Only people with decreased blood flow to the brain, as demonstrated on a PET (positron emission tomographic) scan, are randomized into the COSS study. Among patients randomized into the COSS study, RECON will evaluate whether restoring the blood flow to the brain (with EC-IC bypass surgery) will also improve mental functioning. Participants in both the surgical and medical groups of the COSS study will participate in the RECON study. By comparing the mental functioning of the participants in both treatment groups over the course of 2 years, the investigators hope to determine whether the EC-IC bypass operation also helps improve or maintain mental functioning.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment into Carotid Occlusion Surgery Study

Exclusion Criteria:

* Prior diagnosis of dementia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2004-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cognitive Functioning on Neuropsychological assessment measures | 2 years

SECONDARY OUTCOMES:
Quality of Life and Disability | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Randolph S Marshall, MD, Principal Investigator — Columbia University; Joanne R Festa, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- See also: Click here for more information about this study — http://cosstrial.org/coss/homerecon.asp